CLINICAL TRIAL: NCT05544487
Title: The Effect of Preoperative Factors and Surgical Technique on Postoperative Outcomes in Patients Undergoing Colorectal Resections at South-eastern Europe.
Brief Title: EAST-west Colorectal Study
Acronym: EAST-west
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, George Theodoropoulos, Professor of Surgery, National and Kapodistrian University of Athens
Other Study IDs: EAST-west 2022
Record Dates: First submitted 2022-09-10; First posted 2022-09-16 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Anastomosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colorectal Anastomosis — Differences in intra-operative techniques and surgeon grades

SUMMARY:
Colorectal resection due to benign and malignant diseases is a commonly performed procedure. The continuity of the gastrointestinal tract is re-established by creating an anastomosis. Although such procedures are often performed, anastomotic techniques and postoperative outcomes usually vary. Failure of the anastomosis might be a life-threatening condition after colorectal resection. A relatively high incidence of anastomotic leaks (up to 30%) has been reported worldwide. Anastomotic failure could happen due to several reasons, that are divided into surgeon-related factors and patient-related factors. So far, there has been no data about the incidence of anastomotic leak in the Western Balkans and the Mediterranean countries.The aim of EAST-WEST Colorectal Study 2022 is to investigate differences in patients undergoing colorectal resections, including pre-operative patient preparation, history of prior surgeries and anastomotic techniques. In addition, this study aims to collect data about post-operative complication rate within 30 days post-surgery across Balkan countries (Slovenia, Serbia, Macedonia, Croatia, BIH and Monte Negro), Greece, Romania and Malta, hence the study outcomes could be applicable to the Mediterranean region, in which patients share a common set of characteristics. This would enable variabilities in practice to be identified and differences regarding postoperative outcomes to be highlighted.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-90 years old undergoing colorectal resection with anastomosis due to benign and malignant diseases
* Any of the procedures listed below performed as an emergency or elective surgery, and by any approach; open, laparoscopic or robotic:

  * Right hemicolectomy and extended right hemicolectomy
  * Ileocecal resection
  * Transverse colon resection
  * Segmental colonic resection - i.e. splenic resection
  * Left hemicolectomy
  * Sigmoid resection
  * Rectal resection
  * Pan-proctocolectomy

Exclusion Criteria:

* Closure of ileostomy or colostomy
* Creation of multiple anastomoses
* Small bowel resection
* Pelvic exenteration
* Cytoreductive surgery

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients undergoing colorectal anastomoses due to benign or malignant reasons.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Leakage rate | 30 days

SECONDARY OUTCOMES:
Re-admission rate within the first 30 days post-surgery. | 30 days
30-day postoperative morbidity | 30 days
30-day postoperative mortality | 30 days
Clavien-Dindo complication classification | 30 days
Length of stay | 30 days

IPD SHARING:
Plan to Share IPD: Undecided